CLINICAL TRIAL: NCT03555682
Title: 2-Hydroxybenzylamine: Multiple Dosing Study in Healthy Humans
Brief Title: 2-HOBA: Multiple Dosing Study in Healthy Humans
Acronym: 2-HOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Vanderbilt University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John Rathmacher, PhD, Director of Clinical Research, Metabolic Technologies Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MTI2018-CS01; R44AG055184 (NIH)
Record Dates: First submitted 2018-05-29; First posted 2018-06-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers
Keywords: Multiple Dosage
MeSH Terms: interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a blinded fashion to 2-HOBA or placebo. A computer-generated randomization sequence with a block of size 3 will be used to assign participants at the ratio of 1:2 (placebo:2-HOBA) at each dose level of the treatment. All participants receiving the lower dose regimen will be completed before enrolling participants in the higher dose group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The dietary supplement will be delivered to the Clinical Research Center by the Investigational Pharmacy at Vanderbilt University Medical Center. Staff nurses and participants will be blinded to the capsule content.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- 2-HOBA Low Dose (Experimental): 2-Hydroxybenzylamine acetate: 500mg dose
  Interventions: Dietary Supplement: 2-HOBA
- 2-HOBA High Dose (Experimental): 2-Hydroxybenzylamine acetate: 750mg dose
  Interventions: Dietary Supplement: 2-HOBA

INTERVENTIONS:
Dietary Supplement: 2-HOBA — 2-HOBA is a compound found in buckwheat and is given as 2-HOBA acetate
  Other Names: 2-Hydroxybenzylamine
  Arms: 2-HOBA High Dose; 2-HOBA Low Dose
Dietary Supplement: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to test how well people tolerate a new dietary ingredient called 2-HOBA and how it is metabolized in the body. 2-HOBA is a compound that occurs naturally in buckwheat seeds. This dietary ingredient has been used in animal studies, and single doses have been tolerated well when given to a small group of healthy people. In this study we will test how well people tolerate taking 2-HOBA over 2 weeks and how it is metabolized by the body.

DETAILED DESCRIPTION:
Consenting healthy volunteers between 18 and 59 years old with no morbidity, including males, and females who are not pregnant will be recruited for the study. Eighteen volunteers will be studied with a reasonable sampling of ethnicities from the Nashville area, and an effort will be made to recruit equal numbers of males and females. The study will be conducted by the Vanderbilt Clinical Research Center (CRC).

Based upon single dose pharmacokinetics, two multiple dose regimens will be studied to determine the safety, accumulation kinetics, and pharmacodynamic effects of multiple daily doses administered over 2 weeks. A complete health history and physical examination will be conducted by a physician. An EKG, baseline blood and urine sample, and vital signs will be taken prior to supplement administration. A physician will oversee all clinical aspects of the study and will be responsible for all trial-related medical decisions. Additionally, DNA will be collected from the blood drawn and used to determine if there are any genetic differences in metabolism of 2-HOBA. Volunteers will be given 3 daily doses of either placebo or one of two levels of 2-HOBA to determine the safety, accumulation kinetics, and pharmacodynamic effects of the multiple dose administration over a 2 week period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between 18 and 59 years old;
* Men and women who are not pregnant at the time of study; and
* Not taking any medication 2 weeks prior to or during the study.

Exclusion Criteria:

* Inability to give informed consent;
* Diseases that could manifest symptoms or signs that would confound interpretation of the relationship between 2-HOBA action and potential adverse effects;
* Diseases that could manifest morbidity;
* Known cardiac disease, kidney disease, or hepatic dysfunction;
* Need to discontinue any drug that is administered as standard of care treatment; and
* Unwillingness or inability to use approved birth-control methods.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Multiple Dose Tolerability | 15 Days
  Tolerability will be assessed through adverse event reporting compared with the placebo group (Comparison of number of AE in treated group to number of AE in placebo group).

SECONDARY OUTCOMES:
Measurement of oxidative protein adducts in platelets | 15 Days
  Oxidative protein adducts will be measured in blood platelets as an indication of efficacy (ng adducted protein/mg protein).
Blood Pressure | 15 Days
  Blood pressure will be measured as an indicator of efficacy against oxidative stress (mm Hg).
Maximum Plasma Concentration (Cmax) | Day 1 and Day 15
  Cmax will be calculated from multiple timed plasma measurements (ng/ml).
Area Under the Curve (AUC) | Day 1 and Day 15
  AUC will be calculated from multiple timed plasma measurements (hr*ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pitchford LM, Driver PM, Fuller JC Jr, Akers WS, Abumrad NN, Amarnath V, Milne GL, Chen SC, Ye F, Roberts LJ 2nd, Shoemaker MB, Oates JA, Rathmacher JA, Boutaud O. Safety, tolerability, and pharmacokinetics of repeated oral doses of 2-hydroxybenzylamine acetate in healthy volunteers: a double-blind, randomized, placebo-controlled clinical trial. BMC Pharmacol Toxicol. 2020 Jan 6;21(1):3. doi: 10.1186/s40360-020-0382-y. PMID 31907026